CLINICAL TRIAL: NCT03792308
Title: A Phase 1, Two-part, Double-blind, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of SPR206 in Healthy Volunteers
Brief Title: A First in Human Study of the Safety and Tolerability of Single and Multiple Doses of SPR206 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: Clinical Network Services (CNS) Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR206-101
Record Dates: First submitted 2018-12-17; First posted 2019-01-03 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
Keywords: Safety; Tolerability; Pharmacokinetics; SPR206
MeSH Terms: interventions — Sodium Chloride; Injections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, combined single and multiple ascending dose (SAD and MAD) trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized in a 3:1 ratio of SPR206 to placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPR206 (Experimental): SAD Cohorts: Subjects will receive single doses of SPR206 via IV infusion over one hour. Planned doses to be studied are: 10, 25, 50, 100, 200, 300, 350 and 400mg. If the 300 mg dose is not deemed safe and well-tolerated, a dose of 250 mg will be used.
  MAD Cohorts: Subjects will receive SPR206 via IV infusion over one hour q8h for 7 consecutive days (Cohorts 9 - 12) and over one hour q8h for 14 consecutive days (Cohort 13). Up to five dose groups will be studied. Planned doses will be 25 mg, 50 mg, 100 mg and 150 mg with dosing occurring q8h for 7 consecutive days (Cohorts 9 - 12) and q8h for 14 consecutive days (Cohort 13). Cohort 13 participants will be dosed at a dose deemed safe and tolerable, not to exceed the maximum dose tested in previous MAD dose cohorts.
  .
  Interventions: Drug: SPR206
- Placebo (Placebo Comparator): The placebo used during this study is normal saline (0.9% sodium chloride for injection).
  SAD Cohorts: Subjects will receive single infusions of placebo (0.9% sodium chloride for injection) over one hour.
  MAD Cohorts: Subjects will receive q8h infusions of placebo over 1 hour for 7 consecutive days (Cohorts 9 - 12) and q8h infusions of placebo over 1 hour for 14 consecutive days (Cohort 13).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPR206 — SAD Cohorts: Double-blind dosing will occur in Cohorts 1 - 8. Six participants will receive single doses of SPR206. The dose escalation steps may be altered following review of the safety data upon completion of each cohort.
  MAD Cohorts: Double blind dosing will occur in Cohorts 9 - 13. Six participants in each cohort will receive multiple doses of SPR206. The dose escalation steps may be altered following review of the safety data upon completion of each cohort. Dosing will commence on the morning of Day 1. Three doses will be administered per day at approximately 8 hours apart. Daily dosing will continue for a total of 7 consecutive days for Cohorts 9 - 12 and for a total of 14 consecutive days for Cohort 13.
  Arms: SPR206
Drug: Placebo — 0.9% sodium chloride for injection. SAD Cohorts: Two participants in each cohort will receive matching placebo. MAD Cohorts: Two participants in each cohort will receive matching placebo.
  Other Names: 0.9% sodium chloride for injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of single and multiple intravenous doses of SPR206 when administered to healthy adult volunteers.

DETAILED DESCRIPTION:
This Phase 1 First in Human study is designed to assess the safety, tolerability, and pharmacokinetics of single and multiple intravenous doses of SPR206 when administered to healthy adult volunteers. This is a randomized, double-blind, placebo-controlled, ascending dose, multi-cohort trial. A total of 104 healthy volunteers will be enrolled in 13 cohorts. The study will be conducted in two phases: A single ascending dose (SAD) phase, followed by a multiple ascending dose (MAD) phase. In SAD, participants in Cohorts 1 - 8 will receive one dose of SPR206 or placebo. In MAD, participants in Cohorts 9 - 12 will receive multiple doses of SPR206 or placebo for 7 consecutive days, and a final cohort, Cohort 13, will receive multiple doses of SPR206 or placebo for 14 consecutive days at a dose deemed safe and tolerable and not to exceed the maximum dose administered to participants in Cohorts 9 - 12. In both parts sequential cohorts will be exposed to increasing doses of SPR206.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females (of non-childbearing potential), 18 to 55 years of age (inclusive) at the time of screening.
2. BMI ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive) for all cohorts;
3. Medically healthy without clinically significant abnormalities at the screening visit or Day -1, including:

   1. Physical examination (PE) and vital signs including temperature, pulse, respiratory rate, and blood pressure;
   2. Triplicate electrocardiograms (ECGs) taken at least 1 minute apart with QTcF interval duration less than 450 msec obtained as an average from the triplicate screening and pre-dose Day 1 ECGs after at least 5 min in a semi-supine quiet rest;
   3. Hemoglobin/hematocrit, white blood cell (WBC) count, and platelet count equal to or greater than the lower limit of normal range of the reference laboratory;
   4. Serum creatinine and bilirubin (total and conjugated) equal equal to or less than the upper limit of normal for the reference laboratory. Serum urea, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) equal to or less than 1.5 times the upper limit of normal for the reference laboratory; results of all other clinical chemistry and urine analytes without any clinically significant abnormality.

   Discussion between the PI and the Medical Monitor (MM) is encouraged regarding the potential significance of any laboratory value that is outside of the normal range during the pre-dose period.
4. Be non-smokers (including tobacco, e-cigarettes, nicotine patches, or marijuana) for at least 1 month prior to participation in the study;
5. Willing and able to provide written informed consent;
6. Be willing and able to comply with all study assessments and adhere to the protocol schedule;
7. Have suitable venous access for drug administration and blood sampling;
8. If female, be of non-childbearing potential (e.g. post-menopausal as demonstrated by follicle stimulating hormone (FSH) or surgical sterilization i.e., tubal ligation or hysterectomy). Provision of documentation is not required for female sterilization, verbal confirmation is adequate;
9. If male, a willingness not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, a willingness to use a condom in addition to having the female partner use a highly effective method of birth control (such as an intrauterine device, diaphragm, oral contraceptives, injectable progesterone, subdermal implants, or a tubal ligation). This criterion applies to males (and/or female partners) who are surgically sterile and must be followed from the time of first study drug administration until 90 days after the final administration of study drug.
10. Are fluent in English such that they are able to understand the informed consent form written in English and do not require use of an interpreter.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past three months determined by the PI to be clinically relevant;
2. History of known or suspected Clostridium difficile infection;
3. History of seizure disorders;
4. Positive urine drug/alcohol testing at screening or check-in (Day -1);
5. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C antibodies (HCV);
6. History of substance abuse or alcohol abuse (defined as greater than 2 standard drinks on average each and every day, where 1 standard drink is defined as containing 10 g of alcohol and is equivalent to 1 can or stubby of mid-strength beer, 30 ml nip spirits, or 100 ml wine) within the previous 5 years;
7. Use of any prescription medication or any over-the-counter medication, herbal products, vitamins, diet aids or hormone supplements within 7 days prior to randomisation;
8. Documented hypersensitivity reaction or anaphylaxis to any medication;
9. Donation of blood or plasma within 30 days prior to randomisation, or loss of whole blood of more than 500 mL within 30 days prior to randomisation, or receipt of a blood transfusion within 1 year of study enrollment;
10. Participation in a New Chemical Entity clinical study within the previous 3 months or a marketed drug clinical study within the 30 days before the first dose of IMP. (Washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study);
11. Any other condition or prior therapy, which, in the opinion of the PI, would make the volunteer unsuitable for this study, including unable to cooperate fully with the requirements of the study protocol or likely to be non-compliant with any study requirements.
12. Participants in Cohort 13 should not have participated in any previous cohort of this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events assessments after single and multiple ascending dose administration at baseline and repeatedly until study completion [Safety and Tolerability] | SAD: Up to 7 days; MAD: Up to 21 days for Cohorts 9 - 12 and up to 28 days for Cohort 13.
  This outcome combines the measure of the number of subjects experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatment

SECONDARY OUTCOMES:
Pharmacokinetics: Time to maximum concentration (Tmax) | SAD: Days 1 and 2 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8, 12 and 24 hours post-infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Time to maximum concentration (Tmax) | MAD: Day 1:pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, and 8 hours post morning infusion start. Prior to morning dose on Days 2, 3 and 5 (Cohorts 9 - 12) and prior to morning dose on Days 2, 3, 5, 7, 9, 11, and 13 (Cohort 13).
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Time to maximum concentration (Tmax) | MAD: Day 7 (Cohorts 9 - 12) and Day 14 (Cohort 13) at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8 and 12 hours post morning infusion start. 24, 36, and 48 hours post infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Maximum concentration (Cmax) | SAD: Days 1 and 2 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8, 12 and 24 hours post-infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Maximum concentration (Cmax) | MAD: Day 1 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, and 8 hours post morning infusion start. Prior to morning dose on Days 2, 3, and 5 for Cohorts 9 - 12 and on Days 2, 3, 5, 7, 9, 11, and 13 for Cohort 13.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Maximum concentration (Cmax) | MAD: Day 7 (Cohorts 9 -12) and Day 14 (Cohort 13) at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8 and 12 hours post morning infusion start. 24, 36, and 48 hours post infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Area under the concentration-time curve from time 0 to last measurable time-point (AUC0-t) | SAD: Days 1 and 2 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8, 12 and 24 hours post-infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Area under the concentration-time curve from time 0 to last measurable time-point (AUC0-t) | MAD: Day 1 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, and 8 hours post morning infusion start. Prior to morning dose on Days 2, 3, and 5 (Cohorts 9 - 12) and Days 2, 3, 5, 7, 9, 11, and 13 (Cohort 13).
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Area under the concentration-time curve from time 0 to last measurable time-point (AUC0-t) | MAD: Day 7 (Cohorts 9 - 12) and Day 14 (Cohort 13) at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8 and 12 hours post morning infusion start. 24, 36, and 48 hours post infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | SAD: Days 1 and 2 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8, 12 and 24 hours post-infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | MAD: Day 1 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, and 8 hours post morning infusion start. Prior to morning dose on Days 2, 3, and 5 for Cohorts 9 - 12 and Days 2, 3, 5, 7, 9, 11, and 13 for Cohort 13.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | MAD: Day 7 (Cohorts 9 - 12) and Day 14 (Cohort 13) at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8 and 12 hours post morning infusion start. 24, 36 and 48 hours post infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Terminal Elimination Rate Constant (kel) | SAD: Days 1 and 2 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8, 12 and 24 hours post-infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Terminal Elimination Rate Constant (kel) | MAD: Day 1 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, and 8 hours post morning infusion start. Prior to morning dose on Days 2, 3, and 5 (Cohorts 9 - 12) and Days 2, 3, 5, 7, 9, 11, and 13 (Cohort 13).
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Terminal Elimination Rate Constant (kel) | MAD: Day 7 (Cohorts 9 - 12) and Day 14 (Cohort 13) at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8 and 12 hours post morning infusion start. 24, 36, and 48 hours post infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Terminal half-life (t1/2) | SAD: Days 1 and 2 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8, 12 and 24 hours post-infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Terminal half-life (t1/2) | MAD: Day 1 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, and 8 hours post morning infusion start. Prior to morning dose on Days 2, 3, and 5 (Cohorts 9 - 12) and Days 2, 3, 5, 7, 9, 11, and 13 (Cohort 13).
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Terminal half-life (t1/2) | MAD: Day 1 (Cohorts 9 - 12) and Day 14 (Cohort 13) at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8 and 12 hours post morning infusion start. 24, 36 and 48 hours post infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Terminal clearance (CL) | SAD: Days 1 and 2 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8, 12 and 24 hours post-infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Terminal clearance (CL) | MAD: Day 1 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, and 8 hours post morning infusion start. Prior to morning dose on Days 2, 3, and 5 (Cohorts 9 - 12) and Days 2, 3, 5, 7, 9, 11, and 13 (Cohort 13).
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Terminal clearance (CL) | MAD: Day 7 (Cohorts 9 - 12) and Day 14 (Cohort 13) at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8 and 12 hours post morning infusion start. 24, 36, and 48 hours post infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Volume of distribution (Vd) | SAD: Days 1 and 2 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8, 12 and 24 hours post-infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Volume of distribution (Vd) | MAD: Day 1 at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, and 8 hours post morning infusion start. Prior to morning dose on Days 2, 3, and 5 (Cohorts 9 - 12) and Days 2, 3, 5, 7, 9, 11, and 13 (Cohort 13).
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: Volume of distribution (Vd) | MAD: Day 7 (Cohorts 9 - 12) and Day 14 (Cohort 13) at pre-dose and at 30, 60, 75, 90, 105, 120 and 150 minutes; and 3, 5, 8 and 12 hours post morning infusion start. 24, 36 and 48 hours post infusion start.
  Plasma sample collection for pharmacokinetic analysis
Pharmacokinetics: SPR206 excreted in urine in each collection interval | SAD: Urine samples collected at pre-dose and over the intervals of 0-4 hours, 4-8 hours, 8-12 hours, and 12-24 hours after start of infusion.
  Urine sample collection for measurement of SPR206 excreted in urine over 24 hours.
Pharmacokinetics: SPR206 excreted in urine in each collection interval | MAD: Urine samples collected on Day 1 pre-dose, 0-4 hours and 4-8 hours after start of first infusion. Days 7-8 (Cohorts 9 - 12): 0-4 hours, 4-8 hours, 8-12 hours, 12-24 hours after start of infusion.
  Urine sample collection for measurement of SPR206 excreted in urine over 24 hours.
Pharmacokinetics: SPR206 excreted in urine in each collection interval | MAD: Urine samples collected on Day 1 pre-dose, 0-4 hours and 4-8 hours after start of first infusion. Days 14-15 (Cohort 13): 0-4 hours, 4-8 hours, 8-12 hours, 12-24 hours after start of infusion.
  Urine sample collection for measurement of SPR206 excreted in urine over 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: James Kuo, MBBS, B Med Sci, FRACP, Principal Investigator — Scientia Clinical Research Limited
Locations (1):
- Scientia Clinical Research Ltd., Randwick, New South Wales, Australia

REFERENCES:
- [Derived] Bruss J, Lister T, Gupta VK, Stone E, Morelli L, Lei Y, Melnick D. Single- and Multiple-Ascending-Dose Study of the Safety, Tolerability, and Pharmacokinetics of the Polymyxin Derivative SPR206. Antimicrob Agents Chemother. 2021 Sep 17;65(10):e0073921. doi: 10.1128/AAC.00739-21. Epub 2021 Aug 2. PMID 34339267